CLINICAL TRIAL: NCT00975247
Title: Impact of a Novel Patient Educational Booklet on Colonoscopy Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brennan Spiegel, Associate Professor of Medicine in Residence, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IIR 08-310; Project Number 0013
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Colon Cancer; Colonoscopy
Keywords: Quality Improvement; Colonoscopy; Screening; Colon Cancer; Polyp detection rates; Colonoscopy completion rates; Scope Withdrawal time; Reduce costs through improving bowel prep quality
MeSH Terms: conditions — Colonic Neoplasms | interventions — Quality Improvement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Received Booklet (Active Comparator): Patients who have received colonoscopy preparation booklet
  Interventions: Other: Receiving an educational booklet
- Did not receive booklet (No Intervention): Patients who did not receive colonoscopy preparation booklet

INTERVENTIONS:
Other: Receiving an educational booklet — Patients who receive an educational booklet will be considered to be receiving an intervention
  Other Names: Quality improvement
  Arms: Received Booklet

SUMMARY:
Background: Achievement of colonoscopy outcomes depends on high-quality bowel preparation by patients; yet inadequate preparation is common.

Objective: To develop and test an educational booklet to improve bowel preparation quality.

Design: "Before-and-after" study followed by randomized controlled trial.

Setting: Veteran Affairs medical center.

Patients: Patients undergoing outpatient colonoscopy

Measurements: The investigators first performed cognitive interviews to identify knowledge and belief barriers to high-quality colonoscopy preparation. The investigators then created a patient educational booklet addressing patient barriers to improve preparatory behaviors. The investigators tested the booklet in 2 sequential studies: (1) controlled "before-and-after" study in patients undergoing colonoscopy during 2 consecutive months: 1 without and 1 with the booklet; (2) randomized controlled trial. The outcome in both studies was bowel preparation quality measured on a 6-point Likert scale (>5="good"). In each study the investigators compared the proportion achieving a "good" preparation between groups and performed logistic regression to measure the effect of the booklet on preparation quality while adjusting for the purgative received.

Limitations: Unknown impact on polyp yield and cancer reduction.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled to undergo outpatient colonoscopic CRC screening or surveillance in VAGLA

Exclusion Criteria:

* In patient admissions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Bowel preparation quality, as measured by the Ottawa scale. | 3 years

SECONDARY OUTCOMES:
Adenomatous Polyp Detection | 3 years
Advanced Adenomatous Polyp Detection | 3 years
Cecal Intubation | 3 years
Withdrawal Time | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Brennan MR Spiegel, MD, MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- West Los Angeles VA Healthcare Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Spiegel BM, Talley J, Shekelle P, Agarwal N, Snyder B, Bolus R, Kurzbard N, Chan M, Ho A, Kaneshiro M, Cordasco K, Cohen H. Development and validation of a novel patient educational booklet to enhance colonoscopy preparation. Am J Gastroenterol. 2011 May;106(5):875-83. doi: 10.1038/ajg.2011.75. Epub 2011 Apr 12. PMID 21483463